CLINICAL TRIAL: NCT07102940
Title: Eftilagimod Alpha in Combination With Neoadjuvant Chemotherapy in Patients With Hormone Receptor Positive/HER2-neg Breast Cancer
Brief Title: Efti in Patients With Hormone Receptor Positive/HER2-neg Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Immutep S.A.S. (Industry)
Responsible Party: Principal Investigator, Pavani Chalasani, Professor of Medicine; Director, Division of Hematology Oncology, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAG3-IIT
Record Dates: First submitted 2025-07-02; First posted 2025-08-05 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; HER 2 Negative Breast Cancer; HR Positive/HER-2 Negative Breast Cancer; Stage 1-3
Keywords: breast; cancer; HER2; HR positive
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Efti + NAC Regimens (Experimental): Eftilagimod Alfa (Efti) will be administered subcutaneously at a dose of 30 mg beginning of week 1 of the trial for a total of 3 doses (week 1, 2 and 3). After 3 weeks, efti will be administered starting with week 4, every 2 weeks and combined with either TC or AC.
  NAC regimens:
  * Docetaxel-cyclophosphamide (TC) intravenous (i.v) every 3 weeks (q3w) x 4, or
  * Dose dense Adriamycin-cyclophosphamide (AC) i.v q2w x 4 followed by weekly paclitaxel IV X12 weeks (alternatively weekly nab-paclitaxel can be used per physician's preference if patient unable to tolerate paclitaxel due to infusion reaction). The NAC regimen will be determined by the treating physician prior to starting on this trial.
  Interventions: Drug: Eftilagimod Alfa (Efti); Drug: Docetaxel-cyclophosphamide (TC) intravenous (i.v); Drug: Dose dense Adriamycin-cyclophosphamide (AC) i.v

INTERVENTIONS:
Drug: Eftilagimod Alfa (Efti) — Eftilagimod Alfa (Efti) will be administered subcutaneously at a dose of 30 mg beginning of week 1 of the trial for a total of 3 doses (week 1, 2 and 3). After 3 weeks, efti will be administered starting with week 4, every 2 weeks and combined with either TC or AC
Drug: Docetaxel-cyclophosphamide (TC) intravenous (i.v) — TC will be administered at docetaxel 75mg/m2 IV and cyclophosphamide 600mg/m2 IV every 3 weeks for a total of 4 administrations starting on week 4 of the trial (weeks 4, 7,10, and 13).
  Docetaxel is administered over 60min (dilute in 250 mL NS or D5W to a final concentration of 0.3 to 0.74 mg/mL and administer over 60 minutes).
  Cyclophosphamide is administered over 30-60min (dilute in 250 to 500 mL NS or D5W and administer over 30 to 60 minutes after docetaxel).
  G-CSF support for TC is per institutional SOC guidelines. Efti is to be given always ≥ 30 minutes after TC is finished if both regimens are administered the same day.
Drug: Dose dense Adriamycin-cyclophosphamide (AC) i.v — AC will be administered at doxorubicin 60mg/m2 and cyclophosphamide 600mg/m2 IV every 2 weeks for a total of 4 administrations starting week 4 of the trial (weeks 4, 6, 8 and 10):
  Doxorubicin is administered over 5 min (Dilute with NS to a final concentration of 2 mg/mL and administered as an IV bolus over three to five minutes into a free flowing IV infusion of NS or D5W).
  Cyclophosphamide is administered over 30-60min (Dilute in 250 to 500 mL NS or D5W and administer over 30 to 60 minutes).
  G-CSF support is per SOC/institutional guidelines.
  Paclitaxel is given weekly for a period of 12 weeks (weeks 12 to 23) at 80mg/m2 (Dilute with 250 to 500 mL NS or D5W (final concentration of 0.3 to 1.2 mg/mL) and administered per institutional guidelines). Alternatively nab-paclitaxel weekly can be used (if paclitaxel cannot be used due to allergic reaction).
  Efti is to be given always ≥ 30 minutes after AC or paclitaxel is finished if both regimens are administered the same day.

SUMMARY:
The goal of this interventional study is to determine pathological complete response (pCR) after neoadjuvant chemotherapy (NAC) and Efti treatment. This is a prospective single arm interventional trial in patients with early-stage HR+/HER2 -ve breast cancer (Stage I-III) who are eligible for neoadjuvant chemotherapy (NAC). Enrolled patients will be treated with single agent efti for 3 weeks and then start NAC in combination with efti. There are 2 standard NAC usually used and will be determined by treating physician prior to starting on this trial.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically documented HR+/HER2 neg (defined as ER expression >10% by IHC and/or PR expression > 10% by IHC and HER2 0 or 1+ or 2+ by IHC or FISH ratio <2 or HER2 gene copy number of <6).
* Clinical early-stage breast cancer (Stage I-III) and a candidate for NAC.
* Be informed of the investigational nature of the trial and all pertinent aspects of the trial.
* Have ECOG performance status of 0-2.
* Have the ability to understand and the willingness to sign a written informed -consent document in accordance with institutional and federal guidelines.
* Be ≥ 21 years of age.
* Have serum creatinine < 1.5 x institutional upper limit of normal (IULN) or a calculated creatinine clearance ≥ 30ml/min (calculated by Cockcroft Gault equation), bilirubin ≤ 2.0, and an SGOT/SGPT/alkaline phosphatase ≤ 2.0 x IULN.
* Have adequate bone marrow function (ANC >1000/μL, Platelets >100,000/ml, Hemoglobin >10gm/dL).
* Women of childbearing potential or male patients of reproductive potential with female partners of childbearing potential must not consider getting pregnant and must avoid pregnancy during the trial and for at least 6 months after the last dose of trial treatment. Female and male patients of reproductive potential must practice highly effective methods of contraception with their partners, if of reproductive potential, during treatment and for 6 months following last dose of treatment with IP.

Exclusion Criteria:

* Receiving concurrent anti-neoplastic therapy for another malignancy
* Known documented or suspected hypersensitivity to the components of the trial drug or analogs.
* Stage IV or patients otherwise not indicated for surgery. Patients with oligometastatic disease who are undergoing curative intent treatment are eligible as long as curative intent surgery is planned.
* A woman of child-bearing potential who has a positive serum pregnancy test (within 72 hours) prior to Day 1.
* Breastfeeding
* Serious infection within 4 weeks prior to Day 1 or active acute or chronic infection needing IV antibiotics. Note: Subjects treated for moderately severe infections with oral antibiotics only, may be included, based on consultation with trial Investigator.
* Evidence of severe or uncontrolled cardiac disease within 6 months prior to first dose of trial treatment including: myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI CTCAE version 5.0 Grade ≥ 2, atrial fibrillation > grade 2 not controlled by a pacemaker, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (NYHA III-IV), cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Receives continuous systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days prior to Day 1. Inhaled or topical steroids and physiological replacement doses of up to 10 mg daily prednisone equivalents are permitted in the absence of active auto-immune disease.
* Live vaccine within 30 days of planned Day 1. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Note: non-live vaccines (e.g., non-live influenza vaccine, non-live COVID-19 vaccine) can be given until 3 days prior to planned Day 1.
* Prior anti-LAG-3 therapy (e.g. anti-LAG-3 antibodies).
* Prior high-dose chemotherapy requiring hematopoietic stem cell rescue.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
To determine pathological complete response (pCR) after neoadjuvant chemotherapy (NAC) and Efti treatment | From enrollment to the end of the study (5 years)
  The number of pathological complete responses determined in surgical pathology report. The primary endpoint is pCR to NAC + efti. Simon's 2-stage design will be used. The null hypothesis that the true pCR rate is 0.08 (8%) will be tested against a one-sided alternative. In the first stage, 30 patients will be accrued. If there are 2 or fewer responses in these 30 patients, the study will be stopped. Otherwise, 20 additional patients will be accrued for a total of 50. The null hypothesis will be rejected if 8 or more responses are observed in 50 patients. This design yields a type I error rate of 0.0426 and power of 0.80 when the true pCR rate is 0.20 (20%).

SECONDARY OUTCOMES:
To determine clinical response to Efti + NAC. | From enrollment to the end of study (5 years)
  Clinical response is determined by clinical/imaging measurements of the tumor performed at baseline, during and end of treatment phase.
  Complete clinical response is defined as no measurable disease per imaging and by exam. Partial response is defined as > 15% decrease in baseline measurements by clinical/imaging to complete response criteria (as above) Stable disease is defined as no change in measurements by clinical/imaging +/- 15% . Progressive disease is defined as increase in clinical/imaging measurement by 15% of baseline measurements or development of a new mass/lesion. The % of patients in each response category will be reported as a descriptive measure. .
To determine change in tumor's Ki67 | From enrollment to the end of study (5 years)
  Compare baseline tumor's Ki67 to that in residual tumor after surgical resection. Wilcoxon signed-rank test be done to compare change in Ki67 between 2 specimens for tumors which have residual disease at time of surgery.

IPD SHARING:
Plan to Share IPD: No